CLINICAL TRIAL: NCT03002948
Title: Effect of Clitoris Topography on Orgasm
Brief Title: Effect of Clitoris Location on Orgasm
Acronym: ECTO
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Serdar Aydın, MD, Bezmialem Vakif University
Other Study IDs: ECTO
Record Dates: First submitted 2016-03-24; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low orgasm: Female Sexual Function Index orgasm score below 3.6
  Interventions: Other: Orgasm

INTERVENTIONS:
Other: Orgasm — clitoris volume, suprapubic angle, urethra-levator gap, suburethral triangle area measurement could made using 4 D transperineal ultrasonography. Clitoris fourchette distance, clitoris perineal body distance, clitoris urethra distance could made with special compasses.
  Female Sexual Function Index orgasm domain score

SUMMARY:
Topography and location of clitoris and its parts may affect the orgasm

DETAILED DESCRIPTION:
Orgasm measurement via Orgasm domain of Female Sexual Function Index, clitoris volume, suprapubic angle, urethra-levator gap, suburethral triangle area measurement could made using 4 D transperineal ultrasonography. Clitoris fourchette distance, clitoris perineal body distance, clitoris urethra distance could made with special compasses.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women between 18 and 50 years old
* BMI below 40 kg/m2

Exclusion Criteria:

* BMI over 40 mhg/m2,
* Women younger than 18 years old
* Virgins
* No active sexual intercourse, women with
* Handicapped to get lithotomy position
* Active vulvar and vaginal infection
* Psychiatric diseases
* Drug usage that may cause sexual dysfunction, menopause.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: sexually active women
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
orgasm score | 12 weeks

IPD SHARING:
Plan to Share IPD: No